CLINICAL TRIAL: NCT04262271
Title: A Study to Identify the Prevalence of Device Specific Errors in Inhaler Technique in Adults With Airways Disease
Brief Title: A Study to Identify Errors in Inhaler Technique in Adults
Acronym: SCORES
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/13
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will observe the inhaler technique of people using 13 different inhaler types; record any technique errors being made against checklists developed for each inhaler device based on their manufacturer's guidelines, and reeducate any observed inhaler technique errors as required.

DETAILED DESCRIPTION:
Anyone aged 16 or over who has a lung condition for which they use an inhaler will be invited to join the study. The investigators will recruit a minimum of 650 study participants, with at least 50 participants using each of the 13 inhaler device types selected. These inhaler device types include: Accuhaler, Autohaler, Breezhaler, Easi-breathe, Easyhaler, Ellipta, Genuair, Handihaler, Nexthaler, pMDI, pMDI plus spacer, Respimat and Turbohaler. Participants will be recruited from respiratory outpatient clinics, hospital wards and from staff at Queen Alexandra Hospital (QAH); from integrated outreach lung clinics, GP database searches, clinics run in primary care settings, respiratory support groups in the Hampshire region, and from students at the University of Portsmouth (UoP).

Participants in this study will have their inhaler technique observed and corrected by a specialist clinician, such as a nurse, pharmacist, physiotherapist or doctor using a single-use placebo device. A placebo device is exactly the same as the inhaler that the participant uses, but there is no active medication in the device. If any errors are made using the placebo inhaler, these will be recorded using device-specific checklists based on manufacturers' guidelines.

Correcting inhaler technique is vitally important in the management of respiratory conditions . Observing patients using their inhaler, identifying any errors in their technique, teaching the correct inhaler technique and then observing the patient repeating the procedure correctly should occur at the time of device prescription; however this often does not happen and patients are left unsure how to use their inhaler and errors are commonplace. After inhaler technique has been corrected in this study, a written information sheet with guidance on how to use the inhaler will be provided to each participant to help reinforce the correct technique.

Alongside recording any errors that participants using the inhalers have made, the investigators will also record additional information such as the type of inhaler they are observed using and how long they have been using that inhaler; their age, gender and how many other inhalers they are using in total; which lung condition they have and how badly it affects them and if they have any other medical conditions. The investigators will also record information using a questionnaire called the SPURTM profiling tool, which assesses patients' beliefs and understanding around their medication; this will be done using an iPad/tablet and all data that is inputted will be anonymous and kept securely, as with all other information.

The information collected on this study will help HCP better understand which inhaler technique errors are made most frequently associated with each different inhaler device. The investigators will also use the information gathered in this study, along with additional information gathered from inhaler experts, to develop a method of scoring inhaler technique errors, which will be tested in a future study. Such a scoring system does not currently exist in the UK and will be a valuable tool in clinical practice to accurately measure how good people are at using their inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥16 years
* Have been prescribed (by a doctor or healthcare professional) 1 of 13* inhaler device types for an airways condition.

  *Accuhaler, Autohaler, Breezhaler, Easi-breathe, Easyhaler, Ellipta, Genuair, Handihaler, Nexthaler, pMDI, pMDI plus spacer (e.g. Aerochamber or Volumatic), Respimat and Turbohaler
* Able to provide written informed consent

Exclusion Criteria:

* Currently on treatment with systemic steroids and/or antibiotics for an exacerbation of the participants' airways condition.
* In the opinion of the investigator that the participant will be unable to perform the study procedures

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any person over the age of 16 who uses and inhaler device for an airways condition.
Sampling Method: Non-Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of device-specific inhaler technique errors (ITE), in 13 different devices using manufacturers' guidelines. | one study visit- day 1
  Device Specific inhaler technique errors

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Vos R, Brown T, Longstaff J, Lomax M, Mackenzie H, Hicks A, Rupani H, Gates J, Fox L, Wiffen L, Chauhan AJ. A Study to Investigate the Prevalence of Device-Specific Errors in Inhaler Technique in Adults With Airway Disease (The SCORES Study): Protocol for a Single Visit Prevalence Study. JMIR Res Protoc. 2021 Aug 27;10(8):e26350. doi: 10.2196/26350. PMID 34448728